CLINICAL TRIAL: NCT05132959
Title: The Association Between The Morphometric Parameters of Shoulder and Supraspinatus Tendinosis
Brief Title: The Morphometric Parameters of Shoulder and Supraspinatus Tendinosis
Status: Completed | Type: Observational
Sponsor: Alanya Alaaddin Keykubat University (Other)
Responsible Party: Principal Investigator, Yavuz Yüksel, Assistant professor, Alanya Alaaddin Keykubat University
Other Study IDs: 12-06
Record Dates: First submitted 2021-09-14; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Shoulder Pain; Tendinosis
MeSH Terms: conditions — Shoulder Pain; Tendinopathy | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient Group: Patients with supraspinatus tendinosis
  Interventions: Diagnostic Test: magnetic resonance imaging
- Control Group: Patients without shoulder pain
  Interventions: Diagnostic Test: magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: magnetic resonance imaging — The MRI images of patients who had undergone to shoulder magnetic resonance imaging because of shoulder pain or another pathology were studied

SUMMARY:
Supraspinatus tendinosis one of the most common pathologies of the musculoskeletal system.The aim of this study to investigate the relationship between supraspinatus tendinosis and shoulder morphology with magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
Supraspinatus tendinosis one of the most common pathologies of the musculoskeletal system. It affects 15-50% of the population and its prevalence increases with age. It can lead to useful disability as well as ease of life. Weight, old age and traumas as recurrent risk for SS tendosis. In the literature, there are a large number of small and small numbers among the biology of supraspinologicus tears .The aim of this study to investigate the relationship between supraspinatus tendinosis and shoulder morphology with magnetic resonance imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

* Patients with shoulder pain or healthy controls

Exclusion Criteria:

* Patients with a history of shoulder surgery or trauma, inflammation of the shoulder joint, inflammatory arthritis, space-occupying mass lesions, rupture of the supraspinatus tendon or calcific tendinitis were excluded from the study.

Age Groups: Child, Adult, Older Adult
Study Population: Patients with shoulder pain due to shoulder pathology and another pathology and who have MRI images of the shoulder were recrutied into the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Coracoacromial ligament thickness | three months
  It was measured at the insertion site of the coracoacromial ligament in the lateral part of the acromion
Acromial angle (delta angle) | three months
  It is the angle between the line parallel to the lower face of the acromion and the ground plane
Acromioglenoid angle | three months
  It is the angle between the lower surface of the acromion (a) and the line parallel to the glenoid bone structure
Axial supraspinatus glenoid angle | at the same time
  It is the angle between the supraspinatus fossa (a) and the line parallel to the glenoid bone structure
Coronal supraspinatus glenoid angle | three months
  It is the angle between the line parallel to the supraspinatus fossa and the line parallel to the glenoid bone structure
Acromiohumeral distance | three months
  It is the narrowest distance between the acromion and the humerus
Coracoacromial arch angle | three months
  : It is the angle between the axis of the coracoacromial ligament (running from the coracoid process to the acromion) and the line parallel to the lower surface of the acromion

CONTACTS AND LOCATIONS:
Locations (1):
- Alanya Alaaddin Keykubat University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided